CLINICAL TRIAL: NCT03306017
Title: Study on the Effects of Left Ventricular Assist Device Implantation on the Phenotype of Blood Platelets and Leucocytes
Brief Title: Effects of Left Ventricular Assist Device Implantation on the Phenotype of Blood Platelets and Leucocytes
Acronym: DAV-Hémo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/16/8258; 2016-A01601-50 (Other: ID-RCB)
Record Dates: First submitted 2017-07-24; First posted 2017-10-10 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Cardiac Insufficiency
Keywords: left ventricular assist device; platelet-leukocyte conjugates; lipo-oxygenase products
MeSH Terms: conditions — Heart Failure | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LAVD implantation (Experimental): Ten patients before and after LAVD implantation had blood sampling
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Three venous blood sampling before the left ventricular assist device implantation and 1 and 2 months after implantation in ambulatory patients.

SUMMARY:
To compare in vivo platelet and leukocyte activation and phenotype before and after Left ventricular assist device (LAVD) implantation

DETAILED DESCRIPTION:
The present study plan to investigate platelet activation in vivo using a variety of biomarkers previously identified as sensitive to high shear stress in patients with severe aortic valve stenosis before and after trans arterial valve replacement. As one of the best biomarker is a high degree of platelet-leukocyte interactions, the study will study in parallel leukocytes activation/differentiation. These parameters will be compared at 3 time-points, before and after LAVD implantation in ambulatory patients.

ELIGIBILITY:
Inclusion Criteria:

* elective implantation of LAVD (Heartmate II),
* written informed consent to the study
* Patients with health insurance

Exclusion Criteria:

* treatment or procedure that could affect platelet functions or turn-over(low-dose aspirin is allowed).
* Pregnancy or breastfeeding
* Juridical Protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2019-01-23 (Actual)

PRIMARY OUTCOMES:
Platelet activation | Month 2 after LAVD implantation
  To compare platelet activation in vivo, using a composite criteria determinated by variety of biomarkers of activation analysed by flow cytometry and enzyme-linked immunosorbent assay (ELISA)

SECONDARY OUTCOMES:
Level of circulating platelet-leukocyte conjugate | Month 2 after LAVD implantation
  To determine the level of circulating platelet-leukocyte conjugate by flow cytometry
Changes in leukocyte phenotype | Month 2 after LAVD implantation
  To determine the leukocyte phenotype which is a composite criteria analysed by flow cytometry, ELISA and lipidaemic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Pierre SIE, MD, PhD, Study Chair — University Hospital of Toulouse, Rangueil, Hematology laboratory
Locations (1):
- University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No